CLINICAL TRIAL: NCT06347042
Title: Efficacy of Qigong Exercise on Sleep Quality and Heart Rate Variability in Patients With Fibromyalgia
Brief Title: Effect of Qigong on Sleep Quality in Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Wageih Agwa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/004897
Record Dates: First submitted 2024-02-08; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): receive qigong exercise + routine medical treatment +Anti-inflammatory diet
  Interventions: Other: qigong exercise + routine medical treatment +Anti-inflammatory diet; Other: routine medical treatment +Anti-inflammatory diet only
- control group (Placebo Comparator): receive medical treatment + Anti-inflammatory diet
  Interventions: Other: routine medical treatment +Anti-inflammatory diet only

INTERVENTIONS:
Other: qigong exercise + routine medical treatment +Anti-inflammatory diet — 1. Qigong exercise is from traditional Chinese medicine exercise . Qigong is system coordinating slow-flowing movement, deep rhythmic breathing, and a calm meditative state of min Frequency of exercise 3 days a week and 60 min a day, including a 15 min warm up, 40 min and 5min cool down.
  Arms: study group
Other: routine medical treatment +Anti-inflammatory diet only — 1. Anti-inflammatory diet is characterized by the exclusion of potential inflammatory foods, such as gluten, dairy, free sugar, and ultra-processed food, rich in sugar, hydrogenated fat, and food additives. are some foods with recognized anti-inflammatory potential
  2. routine medical treatment

SUMMARY:
This study aims to determine any significant efficacy of qigong exercise on sleep quality and heart rate variability in patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a disease of unknown and complex an etiopathogenetic, and although pain is its main characteristic, it also stands out for being a disease with multiple symptoms such as fatigue, sleep disorders, anxiety and depressive disorders. For thirty years, various diagnostic criteria, screening and instruments have been developed in the clinical setting, posing a major challenge to researchers and clinicians worldwide. However, the most widely used criterion has been that of the American College of Rheumatology, 1990, as revised in 2016 . The genetic predisposition, environmental triggers and neuromodulation being involved in the onset and course of the disease. The existence of predisposing factors being associated with a high rate of functional disability . FM affects about 5% of the world population. The incidence is higher in women than in men, and the age range in which FM generally appears is between 30 and 35 years. However, FM remains a poorly understood and difficult-to-diagnose condition.

No abnormalities are seen in fibromyalgia in routine clinical laboratory testing or imaging. Functional MRI and other specialized imaging have revealed certain abnormalities in patients with fibromyalgia compared to control subjects.

The subjectivity of the symptoms and the lack of biomarkers, diagnosis is exquisitely clinical, and diagnostic criteria are constantly evolving; early diagnosis and prevention are still elusive goals. Fibromyalgia severity and progression or improvement can be evaluated by means of a plethora of composite tests. Fibromyalgia pathogenesis is not fully understood; hypotheses state that genetic predisposition, stressful life events, peripheral (inflammatory) and central (cognitive-emotional) mechanisms interplay to create pain despeciation owing to neuro-morphological modifications .Treatment should be multimodal and built on four pillars (patient education; fitness; pharmacotherapy; and psychotherapy); the approach should be individualized, symptom-based and stepwise, establishing shared goals with the patient.

Chronic pain and depression exhibit a bidirectional relationship, mediated by neuroplasticity that involves similar brain structures, neurotransmitters, and signaling pathways, leading to both psychological and physical symptoms. Patients with comorbid depression and chronic pain show lower response rates to antidepressants and a higher incidence of suicide attempts than those without chronic pain.

Anxiety and depression are two comorbidities frequently associated with fibromyalgia and chronic pain, being present in 30-50% of patients at the time of disease diagnosis, patients with FM suffer more anxiety and depression than those without the disease . The prevalence of depression in patients with FM is estimated to be between 18 and 36% and between 11.6 and 32.2% for anxiety disorders.

Chronic pain and poor sleep (primary insomnia) provoke persistent stress-immune activation. Given the evidential effects on quality of life and other medical and psychiatric manifestations that chronic pain and insomnia each have, and the notable pain-sleep connections, an exaggerated combined effect .

Poor sleep is reported by almost 80% of patients with fibromyalgia. Epidemiological studies indicate that lower sleep quality is a risk factor for fibromyalgia; poor sleep is strongly and dose-dependently associated with symptom severity in the fibromyalgia population.

Fatigue is widely known and understood, as it is a natural response of the body to some type of physical and mental stress, but it can also be a sign of some possible physical and/or mental disorder, patients with FM report that fatigue is characterized by excessive physical, mental, and cognitive tiredness and that it is usually not alleviated after hours of sleep or rest, which may end up hindering the performance of work or daily tasks, and thus may contribute to the adoption of sedentary behavior . Fatigue is one of the main symptoms reported by patients with FM when asked about the determining factor impacting their overall health, quality of life, and overall perception of this syndrome. Patients with FM have significantly worse levels of quality of life when compared to healthy individuals. So, affecting the socialization, making it difficult for them to work and perform the daily tasks.

Cardiorespiratory fitness evaluation should be considered by general and respiratory physicians /as well as physiotherapists who treat patients diagnosed with fibromyalgia for more accurate diagnosis, exercise prescription and monitoring of patients' status . Heart rate variability biofeedback is a self-management strategy that guides individuals to breathe at a designated resonance frequency of the cardiovascular system. Resonant breathing may reduce FM-related symptoms as well as improve physical functioning and quality of life. Heart rate variability biofeedback for chronic pain, we found no studies testing the feasibility for individuals with FM regarding protocol adherence or acceptability of the treatment.

Current clinical guidelines for the management of patients with FM recommended multimodal conservative treatments to improve the pain-related symptoms, the physical function and the quality of life. Among the conservative treatments, clinical guidelines include non-pharmacological therapies such as exercise therapy, mind-body therapies, patient education, manual therapy, needling therapies, balneotherapy and multimodal therapies Qigong is a mind-body exercise that is similar to tai chi and should be included in future research on mind-body exercises. There is growing evidence Qigong is a modality of traditional Chinese mind-body medicine that has been used to prevent and cure ailments. It is focuses on mind-body integration, is thought to be an effective exercise in promoting physical and mental wellbeing. Core elements of qigong practice involve movements, meditative components, attention to breathing, and promotion of a state of deep relaxation and integration. Qigong, characterized as meditative movement , uses a framework of movement with unique attentional features. A further characterization is as movement-based embodied contemplative practice in which the mind-body , connection is emphasized; qualities and characteristics of movement are distinguished from conventional exercise, and contemplative aspects are considered within a framework of body awareness and somatic approaches.

Qigong is a total body and mind movement that coordinates body posture, movement and breathing . As a mind-body exercise, the key elements of Qigong are body movement, spiritual guidance and controlled breathing, and Qigong can enhance the cardiorespiratory endurance and flexibility of college students, reduce anxiety, alter their state of mind, and improve the psychological well-being, thus promoting the development of their physical and mental health .

Qigong exercise generates an oxygen supply and acid-base balance against the hypoxic effects of underlying pathological conditions. We also propose that Qigong exercise mediated and focused on the local hypoxia environment of tissues might normalize the circulation of metabolic and inflammation accumulation in the tumor tissue and restore the normal metabolism of tissues and cells through calm, relaxation, and extreme Zen-style breathing that gravitates toward preemptive health and medicine. that both tai chi and qigong reduce inflammatory markers, such as C-reactive protein and interleukin-6, displaying a larger pooled effect size than meditation.

Qigong may be effective to improve vital capacity, it is possible to affirm that Qigong is effective in lowering resting heart rate. And in addition to positive comments on core domains that essentially recapitulate the quantitative information (pain, sleep, impact, physical and mental function), health benefits in other areas also are reported (e.g., food allergies, chemical sensitivities, asthma, sleep apnea, migraines, and blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* All patients are female
* Age from 30 to 50 years
* Body mass index (BMI) from 18.5 to 34.9 kg/m2.
* Patients will include if they have been diagnosed with FM by rheumatologists as fulfilling all the ACR criteria (1990, 2011 and 2016)
* All patients are ambulant independently
* Stable medication pattern for at least 2 months.

Exclusion Criteria:

* Presence of any immune diseases or comorbidities that could explain the main symptomatology of FM
* The presence of brain damage, dementia, or neurological disease.
* The presence of psychiatric disorders or current major depressive episode
* Endocrine disorders
* Fractures in upper limb or lower limb
* Participation in regular exercise training of any type in the previous 3 months.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | evaluated beginning and through study completion, an average of8 weeks
  The Pittsburgh Sleep Quality Index (PSQI): It is used to determine self-reported sleep quality and sleep disturbances for the preceding month. It is a consistent and easy for patients and health-care providers in interpreting the indicators of sleep quality. It is a 19-item test and consists of seven components: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) sleep efficiency, (5) sleep disturbance, (6) sleeping medication use and (7) daytime dysfunction. Each component is scored from 0 to 3, and , each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. PSQI (poor sleep: global score > 5
Heart Rate variability | evaluated beginning and through study completion, an average of8 weeks short time 5minutes
  Smart watch-derived HRV provides a practical alternative with excellent accuracy compared with ECG-based HRV for global markers and those characterizing lower frequency components. However, caution is warranted with HRV markers that predominantly assess short-term variability.

SECONDARY OUTCOMES:
Quality of Life o measure the quality of life of patients with problems found fibromyalgia. | evaluated beginning and through study completion, an average of8 weeks
  The FIQR consists of 21 individual questions across three linked domains: function, overall impact and symptoms. All questions pertain to experiences during the past 7 days and are scored using an 11-point numeric rating scale (0 to 10, with 10 denoting the worst possible condition). The function domain contains nine questions addressing activities of daily living .The overall impact domain consists of two questions relating to the overall impact of fibromyalgia on function and overall impact of symptom severity symptoms domain contains 10 questions and evaluates symptoms commonly reported by fibromyalgia. The total FIQR score (out of 100) is the sum of the three modified domain scores, that is: the summed score for the function domain (range 0 to 90, divided by 3), the score for overall impact domain (range 0 to 20) and the score for the symptoms domain (range 0 to 100, divided by 2). scores is classified as mild (≤40), moderate (>40 & ≤63), and severe (>63)
pain self-administered questionnaire | evaluated beginning and through study completion, an average of8 weeks
  is a self-administered or interviewer-administered pain rating scale with four questions related to pain intensity, with responses rated on a numerical rating scale ranging from 0 to 10; "0" is "no pain" and "10" is "pain as bad (excruciating) as you can imagine". Cancer patients rate their worst, least and average pain in the last 24 h and, the pain experienced at the time they were responding to the questionnaire. Pain interference on general activity, mood, walking ability, normal work, relationships with other people, sleep and enjoyment of life were rated on a numerical scale from 0 = "Does not interfere" to 10 = "Interferes completely". The scale comprised of a diagram of a human figure for locating areas of pain and, questions about pain medications and the percentages of pain relief achieved with medications in the last 24 h.
Fatigue :prevalence and severity of fatigue | evaluated beginning and through study completion, an average of8 weeks
  The Fatigue Severity Scale (FSS):one of the most frequently used inventories for measuring fatigue in people with chronic illnesses. The original FSS is a nine-item questionnaire to measure fatigue severity as a unidimensional concept. Some measures are multidimensional and assess several dimensions of fatigue, such as mental and physical fatigue, but the FSS is designed to measure fatigue in a single dimension using the nine items, which represent a single scale. Each FSS item consists of statements that are scored on a seven-point type scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The mean of the nine item scores is used as the FSS score, which ranges from 1 to 7.
Depression and Anxiety assess Depression and Anxiety | evaluated beginning and through study completion, an average of8 weeks
  HADS to assess the levels of anxiety and depression among patients in nonpsychiatric hospital clinics. Items describing somatic symptoms of depression were eliminated from the scale to reduce the effect of physical illness on the depression scores. 14-item self-reporting scale measuring anxiety (7-item subscale) and depression (7-item subscale). Each item is scored on a 4-level Likert type scale ranging from 0 to 3. Mean subscale scores are either normal (0-7), borderline (8-10), or positive for anxiety or depression (11-21). This translates into a maximal score of 21 on each subscale and a total of 42 on the scale

CONTACTS AND LOCATIONS:
Overall Officials: NESSREEN ALNAHAS, Study Director — Department of Physical Therapy for Cardiovascular &Respiratory Disorder and Geriatrics- Faculty of Physical therapy Cairo University
Locations (1):
- Faculty of Physical therapy Cairo University, Cairo, Giza Governorate, Egypt